CLINICAL TRIAL: NCT04966351
Title: Time-restricted Feeding to Mitigate Metabolic Impairments During Circadian Misalignment
Brief Title: Countermeasures to Circadian Misalignment
Acronym: C2CM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: University of Colorado, Denver (Other); Salk Institute for Biological Studies (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19-9666H; R01DK125653 (NIH)
Record Dates: First submitted 2021-05-09; First posted 2021-07-19 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Circadian Rhythm Sleep Disorder of Shift Work Type; Metabolic Disease; Insulin Sensitivity
Keywords: Shift work; Sleep; Blood sugar; Metabolism
MeSH Terms: conditions — Metabolic Diseases; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circadian misalignment (Condition A) (Experimental): Participants will eat meals during the biological nighttime while remaining awake to mimic overnight work shifts.
  Interventions: Behavioral: Circadian Misalignment
- Circadian misalignment with time-restricted feeding (Condition B) (Experimental): Participants will fast during the biological nighttime while remaining awake to mimic overnight work shifts.
  Interventions: Behavioral: Time-restricted feeding; Behavioral: Circadian Misalignment

INTERVENTIONS:
Behavioral: Time-restricted feeding — Each subject will participate in both conditions (CM and CM+TRF)--one in which food is allowed during the nighttime period and one in which food will be restricted to the daytime only. Food intake will be matched across conditions and designed to keep participants weight stable.
  Arms: Circadian misalignment with time-restricted feeding (Condition B)
Behavioral: Circadian Misalignment — Healthy lean subjects will undergo circadian misalignment induced using a simulated night shift-work protocol in both conditions of the study. Each condition will last approximately 6 days.

SUMMARY:
Insufficient sleep and circadian misalignment are independent risk factors for the development of obesity and diabetes, yet few strategies exist to counter metabolic impairments when these behaviors are unavoidable.

This project will examine whether avoiding food intake during the biological night can mitigate the impact of circadian misalignment on metabolic homeostasis in adults during simulated night shift work. Findings from this study could identify a translatable strategy to minimize metabolic diseases in populations that include anyone working nonstandard hours such as police, paramedics, firefighters, military personnel, pilots, doctors and nurses, truck drivers, and individuals with sleep disorders.

DETAILED DESCRIPTION:
People who work evening, night or rotating shifts (i.e. "nonstandard" work hours) represent one in five U.S. employees and are alarmingly 44% more likely to develop Type 2 diabetes (T2D) compared to people who work standard day shifts. Circadian misalignment is one mechanism suggested to increases the risk of obesity and diabetes in people who work non-standard hours, and is highly prevalent and often unavoidable in modern, 24-hour society (e.g. shift work, long work hours, jet lag, medical residency, emergency responders, military personnel, Daylight Savings Time changes, etc). Disruptions in sleep and circadian rhythms have been linked to insulin resistance, increased energy intake, weight gain, and increased total body, abdominal and intrahepatic fat content, yet there have been limited attempts at identifying strategies or countermeasures to prevent the impact of such disruption on T2D risk in a sizeable proportion of the population.

Therefore, the long-term goal is to identify and develop effective, behavioral countermeasures to combat the increased risk for metabolic diseases associated with sleep and circadian disruption when these behaviors are unavoidable. The overall objective for this project is to test the impact of time-restricted feeding to a 7h period in the day as a noninvasive countermeasure to the metabolic impairments associated with circadian misalignment. The central hypothesis is that time-restricted feeding to the daytime period will prevent metabolic impairments during circadian misalignment compared to a condition where energy is consumed throughout the day and night. The rationale for the proposed project is that defining a non-invasive, scalable and feasible countermeasure to circadian misalignment could mitigate the risk of obesity and T2D.

To test the overall hypothesis, a randomized crossover study will be used with a rigorous inpatient diet, activity and light-controlled protocol in healthy men and women. The impact of time restricted feeding during circadian misalignment on metabolic homeostasis will be determined.

Findings from this study represent a critical advancement in the fields of translational circadian and metabolic physiology by identifying and testing a countermeasure to circadian misalignment. Achievement of the proposed aims could lead to the development of new intervention strategies for chronic disease prevention and management. The knowledge to be gained offers the potential to support cost-effective programs that may inform healthcare approach to metabolic disease prevention in populations at risk for these diseases such as shift workers, individuals with sleep disorders and anyone who eats outside of daytime hours.

ELIGIBILITY:
Inclusion Criteria:

1. 18-35 old; men and women; equal numbers of women and men will be included.
2. Body Mass Index (BMI) between 20.0 and 24.9 ("normal" weight).
3. Physical activity history: inactive to habitual moderate physical activity level
4. Sleep/wake history: habitual sleep duration between 7-9.25 hours.
5. Altitude history: Potential subjects must have lived at Denver altitude or higher for at least 3 months prior to inpatient stay.

Exclusion Criteria:

1. Any clinically significant medical, psychiatric, or sleep disorder
2. Use of prescribed medications/supplements/illicit drugs within one month prior to study
3. History of shift work in year prior to study, or travel more than one time zone in three weeks prior to study. [NOTE: Subjects can be studied at a later date.]
4. Women with history of prior gynecological pathology, <1 year post-partum, breast-feeding and/or pregnant.
5. Non-English speakers will be excluded, as we do not have access to a translator who could rely accurate information to the participant for the consent or throughout the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity-derived from glucose tolerance test | Change to be assessed at Day 3, Day 5, Day 31, Day 33.
Muscle tissue lipids-assessed by lipidomic analyses | Change to be assessed at Day 3, Day 5, Day 31, Day 33.

SECONDARY OUTCOMES:
24-hour circulating blood glucose levels-assessed by assay | Change to be assessed at Day 3, Day 5, Day 31, Day 33.
24-hour circulating blood insulin levels-assessed by assay | Change to be assessed at Day 3, Day 5, Day 31, Day 33.
24-hour circulating blood free fatty acid levels-assessed by assay | Change to be assessed at Day 3, Day 5, Day 31, Day 33.

OTHER OUTCOMES:
Cognitive assessments-Karolinska Sleepiness Scale | Change to be assessed at Day 3, Day 5, Day 31, Day 33.
  subjective sleepiness measurement 1-9, 1=Very Alert, 9=Very sleepy, great effort to keep awake, fighting sleep
Cognitive assessments-Positive and Negative Affect Schedule | Change to be assessed at Day 3, Day 5, Day 31, Day 33.
  subjective emotions & feelings, Scores range from 10-50 with higher scores represent higher levels of positive affect of 20 emotions & feelings items, and lower scores represent lower levels of negative affect of 20 emotions & feelings items.
Cognitive assessments- Psychomotor Vigilance Task | Change to be assessed at Day 3, Day 5, Day 31, Day 33.
  reaction time
Cognitive assessments- Conjunction Visual Search Task | Change to be assessed at Day 3, Day 5, Day 31, Day 33.
  reaction time & error rate
Sleep staging-assessed by polysomnography | Change to be assessed at Day 2, Day 4, Day 30, Day 32.
  Electrical activity across the scalp will be measured using polysomnography and sleep will be staged as Wake, Stage 1, Stage 2, Stage 3 and REM.
Sleep quality assessments-assessed by Actiwatch | Change to be assessed at Day 2, Day 4, Day 30, Day 32.
  movement and light sensor equipment
Sleep quality assessments-assessed by Maintenance of Wakefulness Test | Change to be assessed at Day 2, Day 4, Day 30, Day 32.
  onset of sleep latency
Sleep quality assessments-assessed by Leeds Sleep Evaluation Questionnaire | Change to be assessed at Day 2, Day 4, Day 30, Day 32.
  subjective feelings of last night's sleep compared to usual of (1) getting to sleep- (easier, harder), (quicker, slower), (more drowsy, less drowsy); (2) quality of sleep- (more restful, less restful), (few periods of wakefulness, more periods of wakefulness); (3) awakening pattern-(easier, more difficult), (took shorter, took longer); (4) balance and coordination- (less clumsy, more clumsy)
Functional grip strength-measured by hand dynamometer | Change to be assessed at Day 2, Day 4, Day 30, Day 32.
  average force
Functional balance-assessed by multi-sensor recorder | Change to be assessed at Day 1, Day 3, Day 29, Day 31.
  gyroscope, accelerometer, attitude
Systolic and diastolic blood pressure | Change to be assessed at Day 2, Day 4, Day 30, Day 32.
  automatic vitals machine

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Josiane Broussard's Bibliography — http://www.ncbi.nlm.nih.gov/sites/myncbi/1JaM6qKzqsa5p/bibliography/45302103/public/?sort=date&direction=ascending